CLINICAL TRIAL: NCT07365800
Title: The MDK Study: Using a Combination of Methadone-dexmedetomidine-ketamine for Postoperative Pain Control in Patients Undergoing Complex Spine Surgeries.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kiersten Norby, Assistant Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2130514
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spine Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Group receiving the methadone-dexmedetomidine-ketamine medication combination intravenously during anesthesia for complex spine surgery.
  Interventions: Drug: Methadone-dexmedetomidine-ketamine combination
- Routine (No Intervention): Group that receives routine anesthesia with opioid medications during complex spine surgery.

INTERVENTIONS:
Drug: Methadone-dexmedetomidine-ketamine combination — Combination of Methadone-dexmedetomidine-ketamine administered during spine surgery for intra- and post-operative pain management.
  Arms: Intervention

SUMMARY:
This study will investigate whether a combination of three anesthetic medications will reduce intraoperative and postoperative pain in patients undergoing complex spine surgery, and whether it will reduce the use of opioid pain medication after surgery.

DETAILED DESCRIPTION:
Dexmedetomidine, methadone and ketamine offer benefits when used as adjuncts in complex spine surgeries. Dexmedetomidine is reported to attenuate intraoperative stress responses without interfering with neuromonitoring while potentially improving postoperative pain control and reducing opioid consumption in complex spine surgery. Methadone use intraoperatively improves postoperative pain control and reduced opioid requirements following complex spine surgery. Consensus guidelines from the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists support the use of ketamine in acute pain management in surgeries like spine surgery. Perioperative ketamine use in spine surgery results in lower pain scores and reduced opioid utilization postoperatively. The use of dexmedetomidine, methadone and ketamine as adjuncts may improve postoperative pain control while reducing opioid requirements, lowering stress responses, and without significantly impacting neuromonitoring in complex spine surgery or increasing drug related adverse events.

ELIGIBILITY:
Inclusion criteria:

* Age 18-79 years of age
* Patients undergoing complex spine surgery, defined as 3 or more levels
* English-speaking
* Able to consent for themselves

Exclusion criteria:

* Patients who are unable to consent to study participation in English
* Patients who are unable to consent for themselves.
* Patients with prolonged QT syndrome
* Pregnancy

Additional screening measures:

* Preoperative ECG will be performed in preoperative holding as part of standard of care to assess for prolonged QTc prior to administration of methadone as part of SOC.
* Pregnancy test will be performed as part of SOC on the day of surgery.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Effect of the MDK combination during surgery on postoperative opioid consumption | 72 hours postoperatively
  Determine if use of dexmedetomidine, methadone, and ketamine given together intraoperatively has an effect on postoperative opioid consumption following complex spine surgery of 3 or more levels

SECONDARY OUTCOMES:
Effect of MDK combination on overall postoperative pain scores. | 72 hours after surgery
  Determine whether dexmedetomidine, methadone, and ketamine given together intraoperatively has an effect on overall postoperative pain scores following complex spine surgery compared to standard therapy. Pain scores using the visual analog scale, collected by nursing staff during hospital stay, will be used.
Incidence of opioid-related adverse events | 72 hours postoperatively
  Evaluate incidence of opioid related adverse events in patients treated with intraoperative combination of methadone, dexmedetomidine and ketamine compared to standard therapy. The number of adverse events per group will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No